CLINICAL TRIAL: NCT04477980
Title: Retrospective Review on Patients With Culture Negative Empyema
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Honorary Clinical Tutor, Chinese University of Hong Kong
Other Study IDs: CREC 2018.194
Record Dates: First submitted 2020-06-28; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Empyema, Pleural
Keywords: Culture positive empyema; Culture negative empyema; Parapneumonic effusion; Pleural fluid; Pneumonia
MeSH Terms: conditions — Empyema, Pleural; Pneumonia | interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Culture positive empyema: Patients with empyema confirmed by a positive pleural fluid culture, irrespective of its gross fluid appearance
  Interventions: Other: Disease outcome (mortality)
- Culture negative empyema: Patients with empyema confirmed by a gross pus appearance AND a negative pleural fluid culture
  Interventions: Other: Disease outcome (mortality)

INTERVENTIONS:
Other: Disease outcome (mortality) — Mortality rate between the two groups

SUMMARY:
Empyema is associated with a wide range of complication and mortality. It is defined by either a positive pleural fluid culture or grossly pus appearance. However, little is known about the differences in aetiology and outcome between culture-positive empyema (CPE) and culture-negative empyema (CNE). The aim of the current study is to look at the local prevalence of CNE, and compare the clinical outcome between CPE and CNE.

DETAILED DESCRIPTION:
Pneumonia is a common disease and it ranked second as the leading cause of death in Hong Kong in 2016. Among patients suffering from acute pneumonia, up to 57% of them would develop parapneumonic effusion. Without proper treatment, parapneumonic effusion would progress into empyema, which is a clinical emergency. Empyema leads to a longer length of hospital stay, a higher rate of complication and mortality than uncomplicated parapneumonic effusion.

The mainstay of treatment for empyema is antibiotics and drainage. Therefore, identification of causative microorganism is important in guiding the choice of antibiotics. The common bacterial culprits, for community acquired and hospital acquired, were identified by various local and international studies. However, the aetiological agents were still unknown in up to 40% of cases. In addition, the clinical outcomes between culture negative empyema (CNE) and culture positive empyema (CPE) are largely unknown. Data from one Taiwanese study suggested that patients with CPE had a higher in-hospital mortality than those with CNE. However, the primary objective of this study was not putting on the importance of CNE. Therefore, data on outcome of CNE patients remain largely uncertain, either worldwide and local population.

The aim of the current study is to look at the local prevalence of CNE, and compare the clinical outcome between CPE and CNE. Through more understanding of CNE, the clinical management of this patient group may be altered and a better patient outcome is anticipated.

ELIGIBILITY:
Inclusion Criteria:

i. All patients hospitalized for empyema, defined by the presence of purulent pleural fluid or positive culture result from pleural fluid ii. Age greater than 18 years old

Exclusion Criteria:

i. Inappropriate diagnosis of empyema after evaluation ii. Tuberculous pleuritis, defined by presence of Mycobacterium tuberculosis culture from pleural fluid or granulomatous inflammation on pleural biopsy histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A. By using the International Classification of Diseases, Tenth Revision, Clinical Modification code 510.0 or 510.9, all primary hospital discharge diagnosis of empyema during a 5 year period, between 1st January 2013 to 31st December 2018
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Compare the mortality rate within same admission between patients with culture-positive empyema (CPE) and culture-negative empyema (CNE) | Within the same episode of hospitalization or 7 days, whichever longer
  Compare the mortality rate within same admission between patients with culture-positive empyema (CPE) and culture-negative empyema (CNE)

SECONDARY OUTCOMES:
Prevalence of negative pleural fluid culture in patients with empyema | 6 years
  Prevalence of negative pleural fluid culture in patients with empyema
b. Compare other clinical outcomes (length of hospital stay, duration of intravenous antibiotics, number of pleural drainage received, need of surgical treatment, 30-days and 90-days mortality) between patients with CNE and CPE | Within the same episode of hospitalization or 90 days, whichever longer
  Compare other clinical outcomes (length of hospital stay, duration of intravenous antibiotics, number of pleural drainage received, need of surgical treatment, 30-days and 90-days mortality) between patients with CNE and CPE
Investigate the risk factors of failure to obtain culture results in patients with CNE | Within the same episode of hospitalization or 7 days, whichever longer
  Investigate the risk factors of failure to obtain culture results in patients with CNE

CONTACTS AND LOCATIONS:
Overall Officials: Ka Pang Chan, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: upon individual approach for metaanalysis or related study

REFERENCES:
- [Background] Light RW, Girard WM, Jenkinson SG, George RB. Parapneumonic effusions. Am J Med. 1980 Oct;69(4):507-12. doi: 10.1016/0002-9343(80)90460-x. PMID 7424940
- [Background] Chalmers JD, Singanayagam A, Murray MP, Scally C, Fawzi A, Hill AT. Risk factors for complicated parapneumonic effusion and empyema on presentation to hospital with community-acquired pneumonia. Thorax. 2009 Jul;64(7):592-7. doi: 10.1136/thx.2008.105080. Epub 2009 Jan 8. PMID 19131449
- [Background] Taryle DA, Potts DE, Sahn SA. The incidence and clinical correlates of parapneumonic effusions in pneumococcal pneumonia. Chest. 1978 Aug;74(2):170-3. doi: 10.1378/chest.74.2.170. No abstract available. PMID 679746
- [Background] Dean NC, Griffith PP, Sorensen JS, McCauley L, Jones BE, Lee YC. Pleural Effusions at First ED Encounter Predict Worse Clinical Outcomes in Patients With Pneumonia. Chest. 2016 Jun;149(6):1509-15. doi: 10.1016/j.chest.2015.12.027. Epub 2016 Jan 16. PMID 26836918
- [Background] Kim J, Park JS, Cho YJ, Yoon HI, Lee JH, Lee CT, Lim HJ, Kim DK. Predictors of prolonged stay in patients with community-acquired pneumonia and complicated parapneumonic effusion. Respirology. 2016 Jan;21(1):164-71. doi: 10.1111/resp.12658. Epub 2015 Oct 29. PMID 26510382
- [Background] Ferguson AD, Prescott RJ, Selkon JB, Watson D, Swinburn CR. The clinical course and management of thoracic empyema. QJM. 1996 Apr;89(4):285-9. doi: 10.1093/qjmed/89.4.285. PMID 8733515
- [Background] Niederman MS, Mandell LA, Anzueto A, Bass JB, Broughton WA, Campbell GD, Dean N, File T, Fine MJ, Gross PA, Martinez F, Marrie TJ, Plouffe JF, Ramirez J, Sarosi GA, Torres A, Wilson R, Yu VL; American Thoracic Society. Guidelines for the management of adults with community-acquired pneumonia. Diagnosis, assessment of severity, antimicrobial therapy, and prevention. Am J Respir Crit Care Med. 2001 Jun;163(7):1730-54. doi: 10.1164/ajrccm.163.7.at1010. No abstract available. PMID 11401897
- [Background] Tsang KY, Leung WS, Chan VL, Lin AW, Chu CM. Complicated parapneumonic effusion and empyema thoracis: microbiology and predictors of adverse outcomes. Hong Kong Med J. 2007 Jun;13(3):178-86. PMID 17548905
- [Background] Tu CY, Hsu WH, Hsia TC, Chen HJ, Chiu KL, Hang LW, Shih CM. The changing pathogens of complicated parapneumonic effusions or empyemas in a medical intensive care unit. Intensive Care Med. 2006 Apr;32(4):570-6. doi: 10.1007/s00134-005-0064-7. Epub 2006 Feb 15. PMID 16479377
- [Background] Lin YC, Chen HJ, Liu YH, Shih CM, Hsu WH, Tu CY. A 30-month experience of thoracic empyema in a tertiary hospital: emphasis on differing bacteriology and outcome between the medical intensive care unit (MICU) and medical ward. South Med J. 2008 May;101(5):484-9. doi: 10.1097/SMJ.0b013e31816c00fa. PMID 18414163
- [Background] Lindstrom ST, Kolbe J. Community acquired parapneumonic thoracic empyema: predictors of outcome. Respirology. 1999 Jun;4(2):173-9. doi: 10.1046/j.1440-1843.1999.00170.x. PMID 10382237
- [Background] Chen KC, Chen HY, Lin JW, Tseng YT, Kuo SW, Huang PM, Hsu HH, Lee JM, Chen JS, Lai HS. Acute thoracic empyema: clinical characteristics and outcome analysis of video-assisted thoracoscopic surgery. J Formos Med Assoc. 2014 Apr;113(4):210-8. doi: 10.1016/j.jfma.2013.12.010. Epub 2014 Feb 7. PMID 24512757
- See also: assessed on 13th April 2018 — https://www.chp.gov.hk/en/statistics/data/10/27/117.html